CLINICAL TRIAL: NCT04039776
Title: EVALUATION OF BONE PARAMETERS IN PATIENTS WITH PATELLO-FEMORAL DISORDERS WITH TC IN HORTOSTATISM AND CLINOSTATISM: PILOT STUDY
Brief Title: EVALUATION OF BONE PARAMETERS IN PATIENTS WITH PATELLO-FEMORAL DISORDERS
Acronym: FeRo-CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FeRo-CT
Record Dates: First submitted 2019-07-30; First posted 2019-07-31 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Patello Femoral Syndrome
Keywords: CT
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bone patellofemoral joint indices (Experimental): Evaluation of the bone index values in patients affected by patellofemoral joint disorders, obtained from CT scans performed in both orthostatism and clinostatism
  Interventions: Diagnostic Test: "Cone Beam Computed Tomography" (CBCT)

INTERVENTIONS:
Diagnostic Test: "Cone Beam Computed Tomography" (CBCT) — "Cone Beam Computed Tomography "(CBCT), a machine that use a low dose of radiation compared to traditional CT systems, and allows the examination in supine and standing position knee . In this way, for the same patient it will be possible to calculate the bone indexes both in weight-bearing condition and in non-weight-bearing, comparing the values between them, to identify possible differences due to the influence of orthostatism.

SUMMARY:
The aim of the study is to compare, in patients with patellofemoral joint disorders, the values related to the bone indexes of this joint, obtained from CT performed both in orthostatism and clinostatism

DETAILED DESCRIPTION:
The aim of the study is to compare, in patients with patellofemoral joint disorders, the values related to the bone indexes of this joint, obtained from CT performed both in orthostatism and clinostatism.

Young patients with patellofemoral joint pathology, for which a diagnostic examination is necessary in order to determine a possible surgical indication, will be included in this pilot study, and will be evaluated using the "Cone Beam Computed Tomography "(CBCT), a machine that use a low dose of radiation compared to traditional CT systems, and allows the examination in supine and standing position knee . In this way, for the same patient it will be possible to calculate the bone indexes both in weight-bearing condition and in non-weight-bearing, comparing the values between them, to identify possible differences due to the influence of orthostatism.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, between 18 and 50;
2. Pathology or suspected patellofemoral joint pathology in which a CT examination is required for a diagnostic examination;
3. Signature of informed consent.

Exclusion Criteria:

1. Patients incapable of understanding and will;
2. Pregnant women;
3. Patients with history of previous fractures of the knee.
4. BMI> 40.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Distance between tibial tuberosity and trochlear sulcus | 1 month
  It is a direct measure of the valgus alignment

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No